CLINICAL TRIAL: NCT04239456
Title: RehaCom Memory Modules in Moderate-to-severe Traumatic Brain Injury (TBI)
Brief Title: Strategy + RehaCom for Memory Rehabilitation in Traumatic Brain Injury (TBI)
Acronym: REHACOM-NJHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1016-18
Record Dates: First submitted 2019-12-17; First posted 2020-01-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury With Loss of Consciousness
Keywords: TBI; Face memory; Verbal Memory; Learning; Cognition; Memory training; Pilot study; compensatory memory strategies; cognitive rehabilitation

STUDY DESIGN:
Intervention Model Description: This study is a double-blind randomized clinical trial. Participants will be randomly assigned to a treatment group or wait-list control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Group assignments will be concealed and assessments and interventions will be conducted by trained staff blinded to each other's findings and data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Group A (Experimental): Receive intervention 2 weeks after group assignment.
  Interventions: Device: RehaCom (software)
- Group B (Other): Wait List - Receive intervention 3 months after initial testing.
  Interventions: Device: RehaCom (software)

INTERVENTIONS:
Device: RehaCom (software) — RehaCom software has gamified, interactive modules that will help participants practice the application of various memory strategies at custom, increasingly more difficult levels. Instructor will also use the software to teach and demonstrate the use of memory strategies with the domains targeted (i.e., list learning, remembering written/verbal information, and memory for names/faces).

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of "RehaCom," a computerized treatment for memory deficits, in a 16-session, interactive course. Following a manualized approach, the Rehacom modules will be used for the repeated application of the content acquired during 1-on-1 memory strategy training. The goal is to improve face/name, list and verbal memory of patients who survived a moderate to severe traumatic brain injury.

DETAILED DESCRIPTION:
This randomized clinical trial (RCT) consists of 20 chronic moderate-to-severe TBI patients who will receive memory strategy training and complete three memory modules of the RehaCom at one of the Kessler Foundation locations. Changes in attention, processing speed, verbal/non-verbal new learning and memory (NLM) and executive control will be assessed via pre/post and 3-month follow-up assessments before and after the 8-10 week intervention. Self-report questionnaires will also track functional and emotional outcomes such as mood and anxiety, cognition, quality of life, self-efficacy, deficit awareness, community participation, and readiness for occupational functioning

ELIGIBILITY:
Inclusion Criteria:

* Able to read and speak English fluently at the 5th grade level (for testing; software has multilingual support)
* Had a TBI at least 1 year ago
* No history of learning disorders during school years
* Able to use a personal computer (PC) non-stop for 1 hour without health or visual complaints; able to press keyboard buttons.No history of learning disorders

Exclusion Criteria:

* Actively participating in another intervention study
* Distance to Kessler Foundation East Hanover or West Orange location is more than 20 miles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-11-28 (Estimated)

PRIMARY OUTCOMES:
Change in California Verbal Learning Test - II (CVLT-II) performance | Baseline & 10-14 weeks after baseline assessment
  We will use the raw scores for free and cued delayed recall [0-16] where higher scores indicate better verbal recall.
Change in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) - Story Memory performance | baseline & 10-14 weeks after baseline assessment
  Raw scores from Story A and Story B recall [0-50], where higher scores indicate better recall.
Change in Wechsler Memory Scale III - Faces II performance | baseline & 10-14 weeks after baseline assessment
  Delayed Recall Score [0-48] where higher scores indicate better recall.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be available at the individual level except for parties identified by the New Jersey Health Foundation (funding agency) and approved/mandated by the Kessler Foundation Institutional Review Board (IRB).